CLINICAL TRIAL: NCT04103944
Title: A Novel Reconstruction Device for Osteonecrotic Femoral Head Efficacy Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201111037DIB
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Osteonecrosis
Keywords: osteonecrosis; osteonecrotic repair device
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Intervention Model Description: Each patients will be divided into treatment group (osteonecrotic repair device) or control group (core decompression)
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Osteonecrotic Repair Device (Experimental): A biphasic osteochrondral composite method to support the regeneration of articular cartilage in vivo. With its concept that could be securely installed by press-fit without additional fixation, this approach can present an alternative to perform graft harvest and implantation in a single surgery.
  Interventions: Procedure: Osteonecrotic Repair Device
- Core Decompression (Active Comparator): Core decompression is a common surgical procedure that aims to improve vascular inflow by decreasing intraosseous pressure in the femoral head. It is performed that involves removing a cylindrical core of bone from the proximal femur.
  Interventions: Procedure: Core Decompression

INTERVENTIONS:
Procedure: Core Decompression — 10 patients will be randomized chosen in this group
  Arms: Core Decompression
Procedure: Osteonecrotic Repair Device — 10 patients will be randomized chosen in this group
  Arms: Osteonecrotic Repair Device

SUMMARY:
Numerous studies describing surgical treatments to preserve hip replacements has several controversies and none of these procedures are universally accepted nor have compelling evidence for osteonecrosis of the femoral head (ONFH). With developing a newly approach osteonecrotic device surgical procedure to support the regeneration of necrotic bone and articular cartilage in vivo, this will be the first randomized-controlled feasibility study to determine its safety in ONFH patients.

DETAILED DESCRIPTION:
Total of 20 patients were enrolled and randomized in this study. There are two groups, 10 patients in osteonecrotic device group; 10 incore decompression group. After their baseline data has been collected and their surgical procedure has been completed, the following postoperative data collection are then continued to 6 weeks, 12 weeks, 6 months, one year, and two years' prior from the start of their surgery, in order to understand the new approach of the osteonecrotic device's safety in comparison to the core decompression surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally matured between age 20 to 70 (epiphyses of the femoral head are confirmed to be closed on the radiography, CT, or MRI scan
* Patients without any allergies or major systemic or organ diseases
* Patient's affected hip diagnossied as the 3rd stage of ONFH by MRI

Exclusion Criteria:

* Other lower lib fractures
* Pregnancy
* Extensive degenerative arthritis in hip
* Severe osteoporosis in the head and/or neck of the femoral bone
* Rheumatoid immunity or metabolic arthritis that appears to have severe cartilage damage in the hip
* Stiffness in the hip due to other reasons or medical history with its range of motion clinically measures less than 20 degrees in the abduction and less than 90 degrees flexion
* Diagnosed with either Stage 4, 5, or 6, of ONFH classification by either radiography, MR, CT scan.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMAster Universities Osteoartheitis Index (WOMAC) | Baseline before procedure/surgery up to follow up 2 years after
  Questionaire Scoring
Visual Analogue Scale(VAS) | Baseline before procedure/surgery up to follow up 2 years after
  Subjective Pain Scoring
Harris Hip Score (HHS) | Baseline before procedure/surgery up to follow up 2 years after
  Scoring

IPD SHARING:
Plan to Share IPD: No